CLINICAL TRIAL: NCT01862978
Title: Monitoring the Efficacy and Safety of Heparin and Nadroparin in the Acute Phase of Ischemic Stroke
Brief Title: Safety and Efficacy of Heparin and Nadroparin in the Acute Phase of Ischemic Stroke
Acronym: Heparinas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Vladimir Nosal, MD, PhD, Prof.assistant, University Hospital, Martin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTSVKNEUROL001
Record Dates: First submitted 2013-05-20; First posted 2013-05-27 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Heparin; Nadroparin
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Heparin; Nadroparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Heparin (Experimental): Patient receiving Heparin
  Interventions: Drug: Heparin; Drug: Placebo
- Nadroparin (Experimental): Patient receiving nadroparin
  Interventions: Drug: Nadroparin; Drug: Placebo
- Placebo (Placebo Comparator): Patients receiving placebo
  Interventions: Drug: Heparin; Drug: Nadroparin

INTERVENTIONS:
Drug: Heparin
  Arms: Heparin; Placebo
Drug: Nadroparin
  Arms: Nadroparin; Placebo
Drug: Placebo
  Arms: Heparin; Nadroparin

SUMMARY:
The goal of this study is to show the efficacy and safety of heparin and nadroparin in the acute phase of ischemic stroke. Therapeutic agents are administered at intervals of 4.5 to 2 hours after onset of clinical signs. Overall administration of anticoagulant agents will test 72 hours.

Randomized patients will be divided into three groups. The first group of patients will receive heparin intravenously at the beginning of 2500 UI bolus intravenously, followed by intravenous pump 1000 UI / h (18-20 IU / kg / hr) to reach 2-2.5 times the baseline aPTT. After 24 hours, patients will receive the group Nadroparin subcutaneously in the therapeutic dose.

Second group of patients will be administered subcutaneously Nadroparin the therapeutic dose as recommended.

The third group of patients are those who will receive placebo intravenously and 24 hours after receiving nadroparin subcutaneously in the therapeutic dose.

All patients will receive after 24 hours of starting treatment 100 mg of aspirin per orally.

For initiation of treatment will be assessed:

* Modified Rankin Scale, National Institutes of Health Stroke Scale, inclusion, exclusion criteria
* Sign the informed consent and patient randomization
* Laboratory parameters: glucose, creatinine, GGT, K, Na, Cl, blood count, basic coagulation
* Women of childbearing age (pregnancy test)
* History, clinical presentation, medical history, basic internal review of the status (blood pressure, pulse, body temperature, etc.).
* Initial CT examination of the brain
* EKG
* USG sections of extracranial carotid and vertebral arteries
* special hematology factors

If a patient meets all the necessary criteria, he may be given the test substance. During the first 24 hours will be monitored at regular intervals vital functions.

After 24 hours, each patient received subcutaneous Nadroparin the therapeutic dose and also 100 mg of aspirin per orally.

In the interval from 24 to 30 hours of starting treatment the patient will be made:

* Control CT brain
* EKG
* Basic coagulation
* Reduction to stop treatment for newly identified haemorrhage or severe and extensive focal cerebral ischemia by CT scan
* special hematology factors

  72 hours, 7, 30 and 90 days after starting treatment, the patient's clinical evaluation using the Modified Rankin Scale, National Institutes of Health Stroke Scale and Barthel Index.

Safety endpoints: mortality, adverse side effects, bleeding

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke
* female or male gender
* mRS (modified Rankin Scale) 0-1 (min one month before the event)
* NIHSS ≥ 6 and ≤ 25
* Age: 18-80 years
* initiation of therapy in the interval from 4.5 to 24 hours from onset of symptoms of ischemic stroke
* focal neurological deficit of at least 30 min, which was significantly obviously does not disappear before treatment
* patient will participate voluntarily and signed informed consent. Informed consent will be obtained from each patient, guardian or close relative
* patients who are unable to sign, but who are able to understand what means to participate in the study, may give informed consent through eyewitness
* willingness and ability to comply with the protocol

Exclusion Criteria:

* intracranial hemorrhage confirmed by CT scan
* CT image heavy and extensive focal cerebral ischemia
* lacunar syndrome
* epileptic seizure at the beginning of ischemic stroke
* previous or planned treatment with intravenous, intra-arterial thrombolysis, mechanical recanalization or ultrasound assisted thrombolysis
* stroke, myocardial infarction, head trauma in the last 3 months
* tromboctov count below 100 000/mm ³
* therapeutically uncontrolled blood pressure: systolic blood pressure> 185 mmHg or diastolic blood pressure> 110 mmHg
* therapeutically uncontrolled blood glucose ˂ 2.77 or> 22.15 mmol / l
* Known bleeding diathesis, other coagulopathies, severe hepatopathy, severe nephropathy
* patients receiving oral anticoagulants
* current or previous life-threatening bleeding
* major surgery less than 2 weeks ago
* known malignancy
* active TB
* pregnancy
* allergy to Heparin or Fraxiparine
* known alcohol abuse and / or drugs
* active participation in another clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Safety of nadroparine or heparin | DAY 3,7,30,90
  Safety - incidence of intracranial hemorhage
Efficacy of nadroparine or heparin | DAY 3,7, 30, 90
  Efficacy -level of improvement measured by mRS, and NIHSS

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Nosal, MD, PhD, Principal Investigator — Jessenius Faculty of Medicine; Egon Kurca, MD, PhD, prof, Study Director — Jessenius Faculty of Medicine
Locations (1):
- Neurology Clinic Univeristy Hospital in Martin, Martin, Slovakia

REFERENCES:
- [Derived] Dluha J, Sivak S, Kurca E, Dusenka R, Kalmarova K, Turcanova Koprusakova M, Kantorova E, Nosal V. The safety and efficacy of Heparin and Nadroparin compared to placebo in acute ischemic stroke - pilot study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2016 Dec;160(4):543-548. doi: 10.5507/bp.2016.042. Epub 2016 Sep 19. PMID 27646496